CLINICAL TRIAL: NCT00585390
Title: Randomized, Double-Blind, Placebo-Controlled Pilot Trial of Essential Fatty Acid Deficiency Replacement in Early Schizophrenia
Brief Title: Omega-3 Fatty Acid Deficiency Replacement in Early Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Neil Richtand, MD / Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Richtand #1
Record Dates: First submitted 2007-12-28; First posted 2008-01-03 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia; Fatty Acid Deficiency
MeSH Terms: conditions — Schizophrenia | interventions — Fatty Acids, Omega-3; Olive Oil; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Essential omega-3 fatty acid replacement (Experimental)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids; Dietary Supplement: EPA fish oil concentrate; DHA fish oil concentrate
- Placebo (Placebo Comparator)
  Interventions: Other: Olive oil placebo; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — * Essential omega-3 fatty acid replacement therapy with Eicosapentaenoic acid at 3.2 grams
  * Docosahexaenoic acid fish oil concentrate at 1.6 grams
  Other Names: EPA; DHA
  Arms: Essential omega-3 fatty acid replacement
Other: Olive oil placebo — Olive oil capsules, 8 capsules per day
  Other Names: Olive oil
  Arms: Placebo
Dietary Supplement: EPA fish oil concentrate; DHA fish oil concentrate — 3.2 grams for EPA 1.6 grams for DHA
  Other Names: Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA)
  Arms: Essential omega-3 fatty acid replacement
Drug: Placebo — Olive oil capsule
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) that omega-3 fatty acids has on schizophrenia.

DETAILED DESCRIPTION:
The two aims of the study test the hypotheses that correcting omega-3 fatty acid deficiency in the early stages of schizophrenia improves positive symptom treatment response, negative symptom treatment response, and cognition symptom response.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-25 years.
* Diagnosis of MDD and not exhibited symptom remission CDRS-R (> 28 but < 40) despite being administered a standard therapeutic dose of an SSRI continuously for a minimum of 6 weeks.
* Ability and willingness to provide assent and informed, written consent from at least one biological parent.
* Present with biological parent or legal guardian.
* Willingness to maintain current dietary habits.
* Permission from treating physician
* Able to perform fMRI/MRS.

Exclusion Criteria:

* Inability or unwillingness to provide consent.
* Antecedent or concurrent serious medical illness.
* Clinically unstable medical disease, including cardiovascular, hepatic insufficiency, severe renal impairment, gastrointestinal, pulmonary, metabolic, endocrine, obesity or other systemic disease.
* History of seizures, excluding febrile seizures in childhood.
* Patients requiring treatment with any drug which might obscure the action of the study treatment.
* Female patients who are either pregnant or lactating.
* Clinically significant laboratory abnormalities in the last year on CBC or TSH tests.
* Judged clinically to be at suicidal risk (defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within the past 6 months, or a baseline CDRS-R suicide score of >3).
* Hospitalized within the last 3 months
* Greater than 1 year outside appropriate age/grade level
* Pacemaker
* Cerebral aneurysm clip
* Cochlear implant
* Metal fragments lodged within the eye or braces
* Claustrophobia
* Necessity of sedation (no sedation will be given).
* History of loss of consciousness > 10 minutes in duration
* Allergy to seafood.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine positive symptom treatment response in omega-3 fatty acid deficient first-episode schizophrenia patients augmented with omega-3 fatty acid supplementation vs. placebo. | 12 months

SECONDARY OUTCOMES:
Determine negative and cognitive symptom treatment response in omega-3 fatty acid deficient first-episode schizophrenia patients augmented with omega-3 supplementation vs. placebo. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Richtand, MD, Principal Investigator — Unversity of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States